CLINICAL TRIAL: NCT00410592
Title: A Randomized, Open-Label, Comparative 3-Way Crossover Study of 24-Hour Intragastric pH Profile of Once Daily Oral Administration of Esomeprazole 40 mg, Lansoprazole 30 mg, and Pantoprazole 40 mg at Steady State in Hispanic Patients With Symptomatic GERD
Brief Title: Evaluation of 24-Hour Intragastric pH Using Esomeprazole, Lansoprazole, and Pantoprazole in Hispanic Patients With GERD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00106
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; acid reflux; heartburn; PPI; Hispanic
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole; Pantoprazole; Lansoprazole

INTERVENTIONS:
Drug: Esomeprazole 40mg
Drug: Pantoprazole 40mg
Drug: Lansoprazole 30mg

SUMMARY:
This study will be conducted in order to determine safety and efficacy esomeprazole, lansoprazole and pantoprazole control stomach acid by measuring the stomach acid in men and women of Hispanic origin who have GERD.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Males and females ages 18-69 who are of Hispanic origin
* Symptoms of GERD, defined as heartburn at least 2 times a week on average over the last 3 months

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding
* Known intolerance or lack of response to Proton Pump Inhibitors (PPIs) such as Nexium, Prevacid, or Protonix
* Current or relevant history of non-healed ulcers, stomach surgery, or esophageal surgery

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
To compare the pharmacodynamic efficacy in controlling intragastric pH following administration of esomeprazole 40 mg, lansoprazole 30 mg, and pantoprazole 40 mg taken orally, once daily in Hispanic patients with symptomatic GERD.

SECONDARY OUTCOMES:
Compare nocturnal intragastric pH in Hispanic patients with GERD
Compare integrated acidity (IGA) using 24-hour monitoring period among Hispanic patients with GERD
Assess the short-term safety and tolerability of PPIs being studied in Hispanic patients

CONTACTS AND LOCATIONS:
Overall Officials: Marta Illueca, MD, Study Director — AstraZeneca; Kathryn Collison, Study Chair — AstraZeneca
Locations (8):
- United States (7):
  - Research Site, Anaheim, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research SIte, Chapel Hill, North Carolina
  - Research Site, Houston, Texas
- Research Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Morgan D, Pandolfino J, Katz PO, Goldstein JL, Barker PN, Illueca M. Clinical trial: gastric acid suppression in Hispanic adults with symptomatic gastro-oesophageal reflux disease - comparator study of esomeprazole, lansoprazole and pantoprazole. Aliment Pharmacol Ther. 2010 Jul;32(2):200-8. doi: 10.1111/j.1365-2036.2010.04335.x. Epub 2010 Apr 23. PMID 20456300